CLINICAL TRIAL: NCT04130698
Title: Biobehavioral Regulation to Extinguish Smoking While Treating Another Health Risk
Brief Title: Comparing Two Treatments That Both Target Smoking Cessation and Weight Loss at the Same Time.
Acronym: BREATH
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to COVID-19, public health guidelines prevent in-person group meetings.
Sponsor: Rhode Island College (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1819-1483; R15DA045917-01A1 (NIH)
Record Dates: First submitted 2019-10-09; First posted 2019-10-17 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Smoking Cessation; Weight Loss
MeSH Terms: conditions — Smoking Cessation; Weight Loss | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Distress Tolerance (Experimental): Treatment rationale: RAs will explain that there are 3 (not 2 as in the control) key factors that maintain smoking behavior and excess weight: 1) learned habits, 2) the addictive properties of smoking and food, and 3) a way to manage distress. Therefore, to be effective, an intervention designed to simultaneously treat smoking cessation and weight loss must address all 3 key factors. This condition includes both key factors in the control but introduces the third key factor distress tolerance (DT). Toward that end, modules will include: a values discussion; experiential avoidance; distress tolerance; and mindfulness-based ways to manage distress.
  Module 1: Orientation & ACT; Module 2: Avoidance; Module 3: Cognitive Fusion vs. Defusion; Module 4: Self-As-Context; Module 5: Present-Moment-Awareness; and Module 6: Values and Committed Action.
  Interventions: Behavioral: Distress Tolerance; Drug: transdermal nicotine patch
- Active Health Control (Active Comparator): Treatment rationale: RAs will explain that there are 2 key factors that maintain smoking behavior and excess weight: 1) learned habits and 2) the addictive properties of smoking and food. Therefore, to be effective, an intervention designed to simultaneously treat smoking cessation and weight loss must address both key factors. Toward that end, modules will include standard treatment on: the dangers of smoking, excess weight, unhealthy diets and sedentariness; the importance of healthy behaviors; and relaxation exercises to manage stress. These are all key aspects of standard treatment for smoking cessation and weight loss.
  Module 1: Orientation and Health; Module 2: Game Plan; Module 3: Stress and Coping Strategies; Module 4: Physical Activity; Module 5: Changes in Activities, Habits and Lifestyle; and Module 6: Long-Term Rewards.
  Interventions: Drug: transdermal nicotine patch; Behavioral: Active Health Control

INTERVENTIONS:
Behavioral: Distress Tolerance — The group-level intervention is comprised of one 2-hour weekly group sessions with overweight smokers to learn skills and strategies consistent with distress tolerance intervention to quit smoking and lose weight.
  Arms: Distress Tolerance
Drug: transdermal nicotine patch — Participants will use the patch for 8 weeks as outlined by the recommended usage for steps 1-3 going from 21mg for 4 weeks, 14mg for 1 week, and 7mg for 1 week.
  Other Names: the "patch"
Behavioral: Active Health Control — The group-level intervention is comprised of one 2-hour weekly group sessions with overweight smokers to learn skills and strategies consistent with psychoeducation intervention to quit smoking and lose weight.
  Other Names: Psychoeducation
  Arms: Active Health Control

SUMMARY:
The study has two phases. In Phase 1, the investigators will revise and pilot the distress tolerance (DT) protocol that was originally developed and piloted in a previous study (2P20 GM103430, Spas, PI). Despite the 4-week post-intervention treatment outcomes demonstrating the DT protocol's association with smoking cessation and weight loss, several revisions to the DT protocol are important to improve the intervention. First, the investigators will include the overweight/obese smokers' group-level feedback that the investigators collected during the 7-week intervention and at the 4-week post-intervention individual interviews to tailor the DT protocol to meet the unique needs of smokers with excess weight. Subjects from the previous study revealed factors that led to current and/or previous successful smoking cessation and weight loss efforts, barriers to sustaining current and/or previous successful smoking cessation and weight loss efforts, and general feedback about DT intervention for both health risks. The investigators believe revising the DT protocol to include overweight/obese smokers' unique experience with the novel intervention and their acumen about these key factors will improve the intervention and its generalizability to smokers with excess weight. Additional revisions are described elsewhere. After the investigators pilot the revised DT protocol, the investigators will revise the active health control protocol comprised of standard treatment for smoking cessation and weight loss to ensure both protocols equate for intervention contact time. Although both protocols will have some similar content, to avoid any threats to internal validity, no DT-specific material will be included in the control. In Phase 2, the investigators will conduct a two-armed, preliminary randomized controlled trial (RCT) to compare the revised DT protocol's efficacy to the active health control protocol.

DETAILED DESCRIPTION:
In Phase 1, the investigators will revise the distress tolerance (DT) protocol the investigators developed in a previous study. Currently, the DT protocol is comprised of 6 two-hour weekly group sessions. However, based on the data the investigators collected in the previous study, the investigators will revise the DT protocol to have 7 instead of 6 two-hour weekly group sessions. 6 subjects (1 group) will be recruited to pilot the revised DT protocol. All subjects in the pilot will receive the transdermal nicotine patch (TNP). Prior to initiating use of the TNP on quit day, all subjects will be educated about its use and instructed to comply with all the recommended guidelines for usage as outlined in the directions. Smokers who lapse during treatment will be encouraged to set a new quit date and continue to attempt to quit. Subjects who continue to smoke or lapse after quit day will not be instructed to discontinue the patch unless their smoking level reaches 4 cigarettes/day for 4 days. This recommendation is consistent with safe TNP use. Smoking cessation will be objectively verified by expired carbon monoxide levels and saliva cotinine assays. Specifically, subjects who self-report nicotine abstinence will provide an exhaled breath into a Bedfont Micro Smokerlyzer to measure carbon monoxide levels and provide an adequate amount of saliva for cotinine analyses. RAs will wear non-latex gloves and follow all safety protocols for data collection and storage for biochemical materials. the investigators will use an 8ppm cutoff for expired carbon monoxide levels for stated abstinence of 24 hours for 2 weeks and use a cutoff of 10ng/ml for saliva cotinine assays for stated abstinence of 2 weeks or more as cotinine may be incompletely metabolized before this time. Expired carbon monoxide results will be immediately available. Saliva samples will be frozen for shipment to the American Health Foundation (Valhalla, NY) for cotinine level determination by radioimmune assay. Detected values above the stated cutoffs will be considered indicative of smoking. Therefore, smoking cessation and weight loss will be assessed using expired carbon monoxide and weigh-ins during the intervention and saliva cotinine assays and weigh-ins at follow-ups. During Phase 1 post-intervention follow-up, the investigators will revise the active health control protocol comprised of standard treatment for smoking cessation and weight loss to make sure it equates for intervention contact time.

In Phase 2, 48 subjects (8 groups of 6) will be recruited. Both conditions will receive the TNP and follow the protocol previously outlined in Phase 1. Once 6 eligible subjects are recruited, random assignment will be used to determine which of the two treatment conditions the group will receive. We expect to recruit 6 subjects within two weeks, reducing the lag time between a subject's eligibility and starting the intervention. Compensation for subjects' time will also support timely recruitment. To ensure an equal number of groups are assigned to each of the two conditions, assignment will be completed by choosing from among a fixed pool of 8 entries (4 from each condition). Smoking cessation and weight loss outcomes will be assessed using biochemical measures and weigh-ins during the intervention and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* between 18-64 years old
* have been a regular smoker for at least three years
* meet DSM-IV criteria for nicotine dependence
* smoke on average 10 cigarettes per day
* are overweight or obese (25<BMI<40)
* report motivation to quit smoking and lose weight
* speak English.

Exclusion Criteria:

* engaged in a smoking cessation or weight loss intervention
* use medications known to affect smoking cessation or weight loss
* have a medical condition that is a contraindication for transdermal nicotine patch (TNP)
* regularly use other tobacco products
* endorse active suicidal or homicidal ideation
* self-report or meet diagnostic criteria for an alcohol or drug dependence
* self-report or meet diagnostic criteria for an eating or neurocognitive disorder

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
7-day point-prevalence abstinence from smoking | 6-month follow-up assessments from the end of intervention.
  saliva cotinine assays
5% lower weight from baseline. | 6-month follow-up assessments from the end of intervention
  weigh-ins

SECONDARY OUTCOMES:
Include latency to first smoking lapse and latency to smoking relapse | 6-month follow-up assessments from the end of intervention.
  saliva cotinine assays

CONTACTS AND LOCATIONS:
Overall Officials: Jayson J Spas, PhD, MS, Principal Investigator — Associate Professor
Locations (1):
- Rhode Island College, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No